CLINICAL TRIAL: NCT02928731
Title: The Impact of Cancer and Therapy-related Symptoms on Mainland Chinese Children's Physical and Psychological Well-being: An Exploratory Study
Brief Title: Impact of Cancer on the Physical and Psychological Well-being of Children in Mainland China
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: Physical_Mainland
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Child
Keywords: Cancer; Quality of life; Child
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children with cancer: Children met the criteria below were invited to fill in the questionnaires set 1.
  (1) all children should be ages 9-16 years, (2) they should be able to speak and read Chinese, (3) they should have been diagnosed with cancer for at least 2 months and be currently undergoing active treatment, and (4) they should aware of their diseases (cancer).
  Interventions: Other: Questionnaires set 1
- Healthy children: Children met the criteria below were invited to fill in the questionnaires set 2.
  (1) all children should be ages 9-16 years, (2) they should be able to speak and read Chinese, and (3) they should not have cancer or any other chronic illness.
  Interventions: Other: Questionnaires set 2

INTERVENTIONS:
Other: Questionnaires set 1 — Participants were asked to respond to the Chinese version of the Coping Behavior Checklist for Chinese Children, the Chinese University of Hong Kong: Physical Activity Rating for Children and Youth, and the Pediatric Quality of life Inventory: cancer module.
  Groups: Children with cancer
Other: Questionnaires set 2 — Participants were asked to respond to the Chinese version of the Chinese University of Hong Kong: Physical Activity Rating for Children and Youth,and the Pediatric Quality of life Inventory: generic module
  Groups: Healthy children

SUMMARY:
The aim of this study is to explore the impact of cancer and therapy-related symptoms on Mainland Chinese children's physical and psychological well-being.

DETAILED DESCRIPTION:
According to WHO, the annual cancer death has increased to 13 million a year . The cancer incidence of children has also been growing. As the advancement of diagnostic procedure and treatment, the chance of survival has risen considerably over the past decades. The mortality rate of childhood cancer in mainland China has also dramatically decreased during the recent decades.

Nonetheless, the survivors experience low quality of life. When undergoing diagnostic procedures and treatments, children often suffer from multiple symptoms concurrently, such as nausea, fatigue, decreased appetite, pain, and feeling drowsy. These physical symptoms may have long-lasting effects as the treatments last longer. The increase in severity, duration and frequency of physical symptoms may negatively affect recovery of patients in terms of their functional status and positivity, subsequently leading to sadness and anger . Therefore, children will be anxious and stressful when they have cancer. There is considerably evidence to show that children who experience more symptoms have higher levels of depressiveness as well as lower level of physical and psychological functions.

As a matter of fact, studies have found that coping strategies may affect the quality of life. When going through these therapies-related symptoms, children with cancer will feel helpless and have extreme reactions. They may adopt different types of coping strategies, such as screaming, refusing to have treatments or seeking comfort from parents. Some of the strategies may reduce the psychological pressure temporarily, while some other coping strategies can minimize physical pain. All of these may have their impact on quality of life in different degrees. Therefore, recognizing the effect of different coping strategies on both therapy-related symptoms and quality of life is a crucial step to design appropriate interventions that help cancer children to ease treatment related symptoms, improve their quality of life and promote their psychological well-being. On the other hand, a review of the literature has revealed that physical activity is beneficial to cancer patients in terms of their QoL as well as symptom management. Indeed, promoting regular physical activity has been incorporated to rehabilitation guideline for childhood cancer survivors in recent years, so as to enhance both their physical and functional well-beings, as well as, their psychological and emotional well-beings. In fact, the result of a cross-sectional study did show that there is a positive correlation between physical activity level and health-related quality of life . Another study conducted in western country also demonstrated that physical activity level is related to severity of fatigue and health-related quality of life of cancer patients.

Notwithstanding the fact that regular physical activity is beneficial to cancer patients in terms of their psychological health, many children with cancer are recommend not to engage in regular physical activity. They are often advised to take more rest so as to avoid cancer-related or treatment-related fatigue. Given that, it seems also important for us, as health care professionals to examine the physical activity of children hospitalized with cancer before we will be able to design appropriate interventions to promote the adoption and maintenance of regular physical activity, with an ultimate goal to enhance their QoL and psychological well-being.

Although there is compelling evidence to support that therapy-related symptoms, coping strategies and physical activity may have a significant impact on children's quality of life, all of these studies were conducted in western countries, in which, it is hard to reflect the phenomenon in China. On the other hand, notwithstanding the fact that there were several studies conducted in Hong Kong to examine relationship between therapy-related symptoms, coping strategies, physical activity and QoL in cancer children, cultural discrepancies between Hong Kong and China have made applying this finding to be difficult.

this study will explore explore the Impact of Cancer and Therapy-related symptoms on Mainland Chinese Children's Physical and Psychological well-being.

Mainland Chinese hospitalized Children with cancer in the wards of 3 tertiary public hospitals in Beijing will be invited to participate in the study. The pediatric oncology units of these three hospitals will be similar in nature and setting.

The hospitalized children with cancer, who met the inclusion criteria for the study, will be invited to participate. The inclusion criteria are: (1) all children should be ages 9-16 years, (2) they should be able to speak and read Chinese, (3) they should have been diagnosed with cancer for at least 2 months and be currently undergoing active treatment, and (4) they should aware of their diseases (cancer). We excluded children with cognitive and learning problems identified from their medical records.

To compare the impact of therapy-related symptoms on children's quality of life and physical activity level, a group of healthy children having similar standard of living in Mainland China will be invited to participate in the study. The inclusion criteria are: (1) all children should be ages 9-16 years, (2) they should be able to speak and read Chinese, and (3) they should not have cancer or any other chronic illness.

Approval of the study will be obtained from the hospital ethics committees in Mainland China and the University of Hong Kong.

Firstly, the research student will check the eligibility of cancer children by screening their medical records. The research student will then approach the eligible children who are hospitalized in the wards of the pediatric oncology unit. Written consent will be obtained from their parents after they are told about the details of this study. They will be given an option to participate or refuse their child's involvement in the study. In addition, the children who agree to participate will be also invited to put their names on a special child assent form. Both of them will be assured that their participation is totally voluntary and they are allowed to withdraw from the study at any time. After obtaining the participants' demographics from the parents, the children will be asked to complete a set of questionnaires which consists of the Chinese version of Pediatric Quality of life Inventory, Chinese University of Hong Kong: Physical Activity Rating for Children and Youth and Coping Behavior Checklist. About 20 of them will also be selected at random to have a one-to-one, 20 to 30 minutes, semi-structured interview, and all the interviews will be tape-recorded.

Another group of healthy children will be recruited by similar procedures in the community and they will be asked to respond to the same set of questionnaires except the Coping Behavior Checklist.

The independent t-test and chi-square will be used to assess the factors. Descriptive statistics will be used to calculate the mean scores and standard deviation of different scales.

The qualitative data will be analyzed and reported followed by the seven-step analytical procedure of Colaizzi.

ELIGIBILITY:
Inclusion Criteria:

* all children should be ages 9-16 years,
* they should be able to speak and read Chinese,
* they should have been diagnosed with cancer for at least 2 months and be currently undergoing active treatment,
* they should aware of their diseases (cancer).

Exclusion Criteria:

* children with cognitive and learning problems identified from their medical records.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mainland Chinese hospitalized Children with cancer in the wards of 3 tertiary public hospitals in Beijing.
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | baseline
  The quality of life of the participants will be measured by the Pediatric Quality of life Inventory. This instrument consists 27items with 8 subscales。 Items are reverse-scored and linearly transformed into a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) by asking the participants how much of a problem has been experienced over the last month. Participants will be asked to respond to the Chinese version of the Pediatric Quality of Life Inventory at baseline.

SECONDARY OUTCOMES:
Coping strategies used to deal with the cancer and the therapy-related symptoms | baseline
  The Coping strategies of the participants will be measured by the Coping Behavior Checklist for Chinese Children. It started with the question" supposing you were faced with a very stressful event, such as having to go to hospital for surgery, what would you do?" And followed by 8 items. Items 1, 2 and 8 (problem-focused strategies) are scored from 0 to 2 (0 = 'Hardly ever', 1 = 'Sometimes', 2 = 'Often'). Items 3, 4, 5, 6,and 7 (emotional-focused strategy) are scored from 2 to 0 (0 = 'Often', 1 = 'Sometimes', 2 = 'Hardly ever'). The total possible scores range from 0 to 10, and scores of 0 to 3, 4 to 6 and 7 to 10 are interpreted as corresponding to emotional-focused, mixed-focused and problem-focused responses, respectively.Participants will be asked to respond to the Coping Behavior Checklist for Chinese Children at baseline.
Physical activity level | baseline
  The physical activity level of the participants will be measured by The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth. The instrument adopts an 11- point scoring system (0-10) to grade levels of physical activity ranging from no exercise at all (0) to vigorous exercise on most days (10) and taking into consideration the frequency, duration, and intensity of the activity concerned. Accordingly, scores of 0-2, 3-6, and 7-10 are respectively interpreted as low, moderate, and high physical activity levels. Participants will be asked to response to the Chinese University of Hong Kong: Physical Activity Rating for Children and Youth at baseline

CONTACTS AND LOCATIONS:
Overall Officials: William Ho Cheung LI, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No